

# RESEARCH PROTOCOL

#### PARTICULARS OF RESEARCHER

Full Name: Ina Ismiarti binti Shariffuddin

**Title:** Professor Dr

Department: Department of Anaesthesiology, Faculty of Medicine, Universiti Malaya

Office Contact Number: 03-7949 2052

Mobile Number: 012-2353134 Email: ismiarti@ummc.edu.my

Research Expertise: Anaesthesiology, Intensive Care

#### LIST OF CO-RESEARCHERS

#### Prof Dr Rafidah binti Atan

**Department:** Department of Anaesthesiology, Faculty of Medicine, Universiti Malaya

Email: rafidah.atan@ummc.edu.my

# **Associate Prof Dr Chaw Sook Hui**

Department: Department of Anaesthesiology, Faculty of Medicine, Universiti Malaya

Email: sook hui@ummc.edu.my

# Dr Mayura Hanis binti Ahmad Damanhuri

Department: Department of Anaesthesiology, Faculty of Medicine, Universiti Malaya

Email: mayura@ummc.edu.my

# Dr Ngoi Soo Tein

Department: Department of Anaesthesiology, Faculty of Medicine, Universiti Malaya

Email: ngoisootein@um.edu.my

# Dr Tan Kai Ming

Department: Department of Anaesthesiology, Faculty of Medicine, Universiti Malaya

Email: tankaiming@ummc.edu.my

#### RESEARCH PROPOSAL

#### RESEARCH TITLE

Efficacy and Health Economics of Antimicrobial-impregnated Central Venous Catheters (CVCs) compared to Non-impregnated CVCs in Central Line-associated Bloodstream Infection (CLABSI) Prevention in a Malaysia University Hospital Adult Intensive Care Unit (ICU)

**Keywords:** Antimicrobial-impregnated Central Venous Catheters (CVCs), Central Lineassociated Bloodstream Infection (CLABSI), Intensive Care Unit (ICU)

#### 1. INTRODUCTION

Central venous catheters (CVCs) are indispensable in modern critical care as they are highly reliable as intravenous access for administration of vasopressors, inotropes, irritant solutions, total parenteral nutrition and for haemodynamic monitoring. The average central line utilisation ratios in the ICUs across 45 countries were reported at 0.525 (Rosenthal et al., 2021). CVC usage is associated with complications, including central line-associated bloodstream infections (CLABSIs).

The rate of CLABSI is reported at 4.45 per 1000 central line days in ICUs across 45 countries from 2013 – 2018 (Rosenthal et al., 2021). This in turn, is translated to increased healthcare costs and mortality. One of the strategies to reduce the incidence of CLABSI is the use of antimicrobial-impregnated CVCs. These antimicrobial-impregnated CVCs, which can be coated with either antibiotics (e.g. rifampin, minocycline, etc.) or antiseptics (e.g. chlorohexidine, silver sulphadiazine, benzalkonium chloride, etc.) or both, are proposed to be able to reduce the incidence of CLABSI by inhibiting microorganism colonisation on CVCs. A meta-analysis published in 2018 concluded that antimicrobial-impregnated CVCs were significantly effective in reducing CLABSIs and catheter colonisations (Wang et al., 2018). Nevertheless, its efficacy and beneficial effects, particularly in terms of patients' outcome had not been homogenously demonstrated across literature. Moreover, antimicrobial-impregnated CVCs are more expensive compared to non-impregnated ones, and hence its cost-effectiveness remains doubtful.

To date, in our local setting, no study evaluates the efficacy and economic impact of antimicrobial-impregnated CVCs and on patients' outcome. Cost-effectiveness evaluation is important to provide value-based care in clinical practice. This study aims to evaluate the clinical and economic treatment of antimicrobial-impregnated CVCs vs Non-impregnated CVCs in prevention of CLABSI.

# 1.1 Research Questions

1. Is there any difference in central line-associated bloodstream infection (CLABSI) rates between patients using antimicrobial-impregnated central venous catheters (CVCs) and non-impregnated CVCs in Malaysia adult Intensive Care Unit (ICU)?

- 2. Does the use of antimicrobial-impregnated central venous catheters (CVCs) in central line-associated bloodstream infection (CLABSI) prevention in Malaysia adult Intensive Care Unit (ICU) affect patient length of stay when compared to non-impregnated CVCs?
- 3. Does the use of antimicrobial-impregnated central venous catheters (CVCs) in central line-associated bloodstream infection (CLABSI) prevention in the adult Intensive Care Unit (ICU) setting affect healthcare costs when compared to non-impregnated CVCs?
- 4. How antimicrobial resistance features of the bacteria causing central line-associated bloodstream infection (CLABSI) may differ in patients using antimicrobial-impregnated central venous catheters (CVCs) compared to non-impregnated CVCs?

### 2. OBJECTIVES

# **Primary objective:**

• To compare the incidence of central line-associated bloodstream infection (CLABSI) rate in patients using antimicrobial-impregnated central venous catheter (CVCs) and non-impregnated CVCs in Malaysia adult Intensive Care Unit (ICU)

# **Secondary objectives:**

- To determine the length of stay of patients using antimicrobial-impregnated central venous catheter (CVCs) vs non-impregnated CVCs in Malaysia adult Intensive Care Unit (ICU)
- To undertake a cost-effectiveness analysis in prevention of central line-associated bloodstream infection (CLABSI) between patients using antimicrobial-impregnated central venous catheters (CVCs) and non-impregnated CVCs in Malaysia adult Intensive Care Unit (ICU)
- To compare the antimicrobial resistance features of the bacterial species that caused central line-associated bloodstream infection (CLABSI) between patients using antimicrobial-impregnated central venous catheter (CVCs) and that of non-impregnated CVCs in Malaysia adult Intensive Care Unit (ICU)

#### 3. METHODOLOGY

#### 3.1 Study Location

The study will be conducted in the adult Intensive Care Unit (ICU) of Universiti Malaya Medical Centre (UMMC), which is a mixed medical/surgical ICU.

# 3.2 Study Period

The study will be conducted over a period of one year.

# 3.3 Study Design

The study will be conducted as a randomised-controlled trial.

# 3.4 Study Population

#### Inclusion criteria:

- Patients aged 18 years old and above who are admitted to the ICU of UMMC during the study period
- Patients who require a CVC during ICU stay

#### **Exclusion Criteria:**

- Patients who refuse to participate in the study
- Patients with known hypersensitivity reaction to CVC materials
- Patients with pre-existing diagnosis of central line-associated bloodstream infection (CLABSI) upon admission to the ICU
- Patients with pre-existing bloodstream infection upon admission to the ICU
- Patients with a pre-existing CVC, where sterility during placement may be compromised (e.g. in an emergency situation)
- Patients with indwelling CVC less than 48 hours
- Patients who had poor compliance to catheter bundle care during CVC handling throughout the indwelling catheter period
- Patients who require > 1 CVC or other central venous access

# 3.5 Sampling Method

All adult patients who require a CVC insertion as part of their standard routine treatment in ICU will be recruited. After the recruitment, the patients will be randomly assigned to one of the two different groups using a computer: control group who receives non-impregnated CVC and investigational group who receives antimicrobial-impregnated CVC.

# 3.6 Sample Size

Our local data at ICU, UMMC reported the incidence of CLABSI per 1000 catheter days in the first 6 months of 2022, to be 12.18. Using SAS® for sample size calculation, in order to detect a clinically significant reduction of CLABSI by 30%, and assuming a two-sided type I error protection of 0.05 and a power of 0.80, we calculated a sample size of 50 patients is required. To incorporate a 10% drop out rate, we therefore aim to recruit 55 patients in each arm (antimicrobial-impregnated CVCs, n=55; non-impregnated CVCs, n=55). This will make up to a total sample size of 110.

# 3.7 Variables/ Parameters

# 3.7.1 Dependent Variables

# 3.7.1.1 Primary Outcome

The primary outcome investigated is the central line-associated bloodstream infection (CLABSI) rate, expressed in cases per 1000 catheter days. The diagnosis of CLABSI will be based on the CDC-NHSN definition.

# 3.7.1.2 Secondary Outcomes

The secondary outcomes investigated included:

- i. ICU Length of stay of patients diagnosed with CLABSI
- ii. Healthcare costs of patients diagnosed with CLABSI
- iii. Antimicrobial resistance profiles of the bacterial species isolated from patients diagnosed with CLABSI

#### 3.7.2 Other Parameters

Baseline patient data will be included as concomitant study parameters. Relevant patient and clinical data including basic demographic information (age, gender, and ethnicity), known underlying diseases, previous antibiotic exposure within 90 days, and admission date will be extracted from the clinical database for correlation and risk factor analyses.

For patients diagnosed with CLABSI, information including the number of days a patient spent in the hospital prior to strain isolation, number of days and type(s) of antibiotics used in said patient, hospital-generated antibiograms for each strain, patient risk factors for nosocomial infection associated with an isolate, previous surgeries or hospitalizations of the patient prior to isolation, location of a patient within the hospital prior to strain isolation and ICU admission, and any other information pertinent to a specific strain that will not identify a patient will be collected.

# 3.8 Data Collection

# 3.8.1 Clinical and patient data collection

A form comprising all study parameters will be prepared for data recording and collection. The data will be collected and handled confidentially by the investigators.

# 3.8.2 Bacterial strains collection and molecular assays

For patients who develop CLABSI during their ICU stay, routine blood culture will be obtained and processed at the Medical Microbiology Diagnostic Laboratory, UMMC to identify the bacterial species. Bacterial species identification and antimicrobial susceptibility testing will be conducted using an automated VITEK 2 system (bioMerieux, Marcy-l'Etoile, France), according to standardized protocols. All bacterial strains will be transported to the bacteriology research laboratory at the Department of Medical Microbiology, Faculty of Medicine, UM for further molecular analyses. Polymerase chain reaction (PCR) assays will be conducted to further confirm the identity and genotypes of the bacterial isolates and to determine the antimicrobial resistance-conferring genes that corresponded to the antimicrobial resistance phenotypes of the isolates. Established primer sequences from previous studies will be adapted and PCR assays will be performed using optimized laboratory protocols (Ngoi et al., 2021; Muhamad et al., unpublished data). No additional biological samples will be taken in addition to routine practice and no additional invasive procedures will be performed on the study participants. Hence, there will be no added potential harm to the study participants. The costs for further molecular analyses will be covered by the grant and will not be borne by the patients.

# 3.9 Data Analysis

The data will be analysed using the SPSS Software. Descriptive statistics will be expressed as percentages unless otherwise stated. Categorical variables will be expressed as percentages and compared using the Chi-square or Fisher's exact test, whichever is appropriate. Variables with a univariate test value of less than 0.05 (p-value) will be included in a multivariate analysis using a logistic regression model. Odds ratios (OR) and 95% confidence intervals (CI) will be calculated to identify the risk factors associated with the development of CLABSI in patients. In all instances, a p-value of less than or equal to 0.05 will be considered significant.

#### **FUNDING**

This study will be funded by Teleflex Research Grant (RM50000).

#### RESEARCH DATA MANAGEMENT

All data collected will be handled confidentially according to the Good Clinical Practice Guidelines. The paper case report forms will be stored within a locked cabinet at the Department of Anaesthesiology, Faculty of Medicine, Universiti Malaya. The electronic case report forms will be kept in a password-protected laptop. Only the study investigators will have access to the research data. The data will be kept for seven years upon completion of study. The results of the study will be reported in a thesis. The results will also be presented in conferences and published in scientific journals.

### POTENTIAL RESEARCH IMPACT

The usage of antimicrobial-impregnated central venous catheters (CVCs) among adult critically ill patient in the Intensive Care Unit (ICU) can reduce central line-associated bloodstream infections (CLABSIs) and this will translate to reduced patients' length of stay and healthcare costs.

# **GANTT CHART**

| | 2023 | | | | | | | | | | 2024 | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Research Activities | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 |
| Ethics submission | | | | | | | | | | | | | | | | | | | | | | |
| Patient recruitment | | | | | | | | | | | | | | | | | | | | | | |
| Data collection | | | | | | | | | | | | | | | | | | | | | | |
| Data analysis | | | | | | | | | | | | | | | | | | | | | | |
| Completion and submission of manuscript | | | | | | | | | | | | | | | | | | | | | | |
| Publication and scientific presentations | | | | | | | | | | | | | | | | | | | | | | |

#### REFERENCES

- Alotaibi, N. H., Barri, A., & Elahi, M. A. (2020). Length of Stay in Patients With Central Line-Associated Bloodstream Infection at a Tertiary Hospital in the Kingdom of Saudi Arabia. *Cureus*, *12*(10). https://doi.org/10.7759/CUREUS.10820
- Atilla, A., Doğanay, Z., Kefeli Çelik, H., Demirağ, M. D., & Kiliç, S. S. (2017). Central line-associated blood stream infections: characteristics and risk factors for mortality over a 5.5-year period. *Turkish Journal of Medical Sciences*, 47(2), 646–652. https://doi.org/10.3906/SAG-1511-29
- Benenson, S., Cohen, M. J., Schwartz, C., Revva, M., Moses, A. E., & Levin, P. D. (2020). Is it financially beneficial for hospitals to prevent nosocomial infections? *BMC Health Services Research*, 20(1), 1–9. https://doi.org/10.1186/S12913-020-05428-7/TABLES/5
- Bloodstream Infection (BSI) Events (Central Line-Associated Bloodstream Infection (CLABSI) and non-central line-associated Bloodstream Infection) Protocols. (2022, January). Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network (NHSN). https://www.cdc.gov/nhsn/psc/bsi/
- Cai, Y., Zhu, M., Sun, W., Cao, X., & Wu, H. (2018). Study on the cost attributable to central venous catheter-related bloodstream infection and its influencing factors in a tertiary hospital in China. *Health and Quality of Life Outcomes*, 16(1). https://doi.org/10.1186/S12955-018-1027-3
- Chen, Y. M., Dai, A. P., Shi, Y., Liu, Z. J., Gong, M. F., & Yin, X. B. (2014). Effectiveness of silver-impregnated central venous catheters for preventing catheter-related blood stream infections: a meta-analysis. *International Journal of Infectious Diseases: IJID: Official Publication of the International Society for Infectious Diseases*, 29, e279–e286. https://doi.org/10.1016/J.IJID.2014.09.018
- Chong, H. Y., Lai, N. M., Apisarnthanarak, A., & Chaiyakunapruk, N. (2017). Comparative efficacy of antimicrobial central venous catheters in reducing catheter-related bloodstream infections in adults: Abridged cochrane systematic review and network meta-analysis. *Clinical Infectious Diseases*, 64, S131–S140. https://doi.org/10.1093/cid/cix019
- Current HAI Progress Report 2020 National and State Healthcare-Associated Infections Progress Report | HAI | CDC. (2021, October). https://www.cdc.gov/hai/data/portal/progress-report.html
- Dal Forno, C. B., Correa, L., Scatena, P. D., Silva, C. V., Shiramizo, S., Pavão dos Santos, O. F., Cendoroglo Neto, M., Teich, V., Teich, N., & Sardenberg, C. (2012). Bloodstream Infection in the Intensive Care Unit: Preventable Adverse Events and Cost Savings. *Value in Health Regional Issues*, 1(2), 136–141. https://doi.org/10.1016/J.VHRI.2012.10.002
- Dey, S., Tarat, A., Bhattacharyya, R., & Saikia, L. (2021). Demographic characteristics and microbial profile of central line associated blood stream infections in the central intensive care unit. *International Journal of Medical and Health Research*, 7(7), 49–52. https://www.researchgate.net/publication/353715961

- Dube, W. C., Jacob, J. T., Zheng, Z., Huang, Y., Robichaux, C., Steinberg, J. P., & Fridkin, S. K. (2020). Comparison of Rates of Central Line-Associated Bloodstream Infections in Patients With 1 vs 2 Central Venous Catheters. *JAMA Network Open*, 3(3). https://doi.org/10.1001/JAMANETWORKOPEN.2020.0396
- Gershengorn, H. B., Garland, A., Kramer, A., Scales, D. C., Rubenfeld, G., & Wunsch, H. (2014). Variation of Arterial and Central Venous Catheter Use in United States Intensive Care Units. *Anesthesiology*, 120(3), 650–664. https://doi.org/10.1097/ALN.0000000000000000
- Gopal Katherason, S., Naing, L., Jaalam, K., Kamarul Imran Musa, K., Nik Abdullah, N. M., Aiyar, S., Bhojwani, K., Harussani, N., Abdul Rahman, A., & Ismail, A. (2010). Prospective surveillance of nosocomial device-associated bacteremia in three adult intensive units in Malaysia. *Tropical Biomedicine*, 27(2), 308–316. http://mymedr.afpm.org.my/publications/21817
- Krikava, I., Kolar, M., Garajova, B., Balik, T., Sevcikova, A., Roschke, I., & Sevcik, P. (2020). The efficacy of a non-leaching antibacterial central venous catheter a prospective, randomized, double-blind study. *Biomedical Papers*, *164*(2), 154–160. https://doi.org/10.5507/BP.2019.022
- Lai, N. M., Chaiyakunapruk, N., Lai, N. A., O'Riordan, E., Pau, W. S. C., & Saint, S. (2016). Catheter impregnation, coating or bonding for reducing central venous catheter-related infections in adults. In *Cochrane Database of Systematic Reviews* (Vol. 2016, Issue 3). John Wiley and Sons Ltd. https://doi.org/10.1002/14651858.CD007878.pub3
- Leistner, R., Hirsemann, E., Bloch, A., Gastmeier, P., & Geffers, C. (2013). Costs and prolonged length of stay of central venous catheter-associated bloodstream infections (CVC BSI): a matched prospective cohort study. *Infection 2013 42:1*, 42(1), 31–36. https://doi.org/10.1007/S15010-013-0494-Z
- Lin, F. F., Murphy, N., Martinez, A., & Marshall, A. (2022). An audit of central venous catheter insertion and management practices in an Australian tertiary intensive care unit: A quality improvement project. *Intensive and Critical Care Nursing*, 103217. https://doi.org/10.1016/J.ICCN.2022.103217
- Lin, K. Y., Cheng, A., Chang, Y. C., Hung, M. C., Wang, J. T., Sheng, W. H., Hseuh, P. R., Chen, Y. C., & Chang, S. C. (2017). Central line-associated bloodstream infections among critically-ill patients in the era of bundle care. *Journal of Microbiology, Immunology, and Infection = Wei Mian Yu Gan Ran Za Zhi*, 50(3), 339–348. https://doi.org/10.1016/J.JMII.2015.07.001
- Lorente, L., Lecuona, M., Jiménez, A., Lorenzo, L., Diosdado, S., Marca, L., & Mora, M. L. (2014). Cost/benefit analysis of chlorhexidine-silver sulfadiazine-impregnated venous catheters for femoral access. *American Journal of Infection Control*, 42(10), 1130–1132. https://doi.org/10.1016/J.AJIC.2014.06.027
- Lorente, L., Lecuona, M., Jiménez, A., Lorenzo, L., Santacreu, R., Ramos, S., Hurtado, E., Buitrago, M., & Mora, M. L. (2015). Efficiency of chlorhexidine-silver sulfadiazine-impregnated venous catheters at subclavian sites. *American Journal of Infection Control*, 43(7), 711–714. https://doi.org/10.1016/J.AJIC.2015.03.019

- Lorente, L., Lecuona, M., Jiménez, A., Santacreu, R., Raja, L., Gonzalez, O., & Mora, M. L. (2014). Chlorhexidine-silver sulfadiazine-impregnated venous catheters save costs. *American Journal of Infection Control*, 42(3), 321–324. https://doi.org/10.1016/J.AJIC.2013.09.022
- Mermel, L. A., Allon, M., Bouza, E., Craven, D. E., Flynn, P., O'Grady, N. P., Raad, I. I., Rijnders, B. J. A., Sherertz, R. J., & Warren, D. K. (2009). Clinical Practice Guidelines for the Diagnosis and Management of Intravascular Catheter-Related Infection: 2009 Update by the Infectious Diseases Society of America. In *Clinical Infectious Diseases* (Vol. 49, Issue 1, pp. 1–45). https://doi.org/10.1086/599376
- Mishra, S. B., Misra, R., Azim, A., Baronia, A. K., Prasad, K. N., Dhole, T. N., Gurjar, M., Singh, R. K., & Poddar, B. (2017). Incidence, risk factors and associated mortality of central line-associated bloodstream infections at an intensive care unit in northern India. *International Journal for Quality in Health Care*, 29(1), 63–67. https://doi.org/10.1093/INTQHC/MZW144
- Muhamad, A. N., Ngoi, S. T., Teh, C. S. J., Draman, M. R., Adnan, Y. K., Tan, S. C., Abbas, A. A., Tang, S. N., Karunakaran, R., Kukreja, A., Mohamad Razali, S. Z., Hontz, R. D., Gregory, M. J., & Ponnampalavanar S. (2022). The incidence and microbial characteristics of surgical site infections following traumatic orthopaedic surgeries in a tertiary hospital in Malaysia. (Unpublished data)
- Nakamura, I., Fukushima, S., Hayakawa, T., Sekiya, K., & Matsumoto, T. (2015). The additional costs of catheter-related bloodstream infections in intensive care units. *American Journal of Infection Control*, *43*(10), 1046–1049. https://doi.org/10.1016/J.AJIC.2015.05.022
- Ngoi, S. T., Chong, C. W., Ponnampalavanar, S. S. L. S., Tang, S. N., Idris, N., Abdul Jabar, K., Gregory, M. J., Husain, T., & Teh, C. S. J. (2021). Genetic mechanisms and correlated risk factors of antimicrobial-resistant ESKAPEE pathogens isolated in a tertiary hospital in Malaysia. *Antimicrobial Resistance & Infection Control*, 10(1), 70. https://doi.org/10.1186/s13756-021-00936-5
- Novosad, S. A., Fike, L., Dudeck, M. A., Allen-Bridson, K., Edwards, J. R., Edens, C., Sinkowitz-Cochran, R., Powell, K., & Kuhar, D. (2020). Pathogens causing central-lineassociated bloodstream infections in acute-care hospitals-United States, 2011-2017. *Infection Control and Hospital Epidemiology*, 41(3), 313–319. https://doi.org/10.1017/ICE.2019.303
- Pandit, P., Sahni, A. K., Grover, N., Dudhat, V., Das, N. K., & Biswas, A. K. (2021). Catheter-related blood stream infections: prevalence, risk factors and antimicrobial resistance pattern. *Medical Journal Armed Forces India*, 77(1), 38–45. https://doi.org/10.1016/J.MJAFI.2019.07.002
- Pepin, C. S., Thom, K. A., Sorkin, J. D., Leekha, S., Masnick, M., Preas, M. A., Pineles, L., & Harris, A. D. (2015). Risk factors for central-line-associated bloodstream infections: a focus on comorbid conditions. *Infection Control and Hospital Epidemiology*, 36(4), 479–481. https://doi.org/10.1017/ICE.2014.81

- Polderman, K. H., & Girbes, A. R. J. (2002). Central venous catheter use: Part 2: Infectious complications. In *Intensive Care Medicine* (Vol. 28, Issue 1, pp. 18–28). https://doi.org/10.1007/s00134-001-1156-7
- Preventing Central Line-Associated Bloodstream Infections: A Global Challenge, A Global Perspective. (2012). https://www.jointcommission.org/resources/patient-safety-topics/infection-prevention-and-control/central-line-associated-bloodstream-infections-toolkit-and-monograph/
- Rai, V., Yuet-Meng, C., Rosenthal, V. D., Hasan, S., Zaman, K., Mansor, M., Sri, S., Sri Ponnampala, L., Shiham, A., Abidin, Z., Manikavasagam, J., Phuong, M., Binh, G., O E Le N E Lim, M D ', J., Auzani Othman, A., Ling, S., Seng Gan, M D ', C., Aziz, A., Latif, H. A., ... Mohamad Yusof, B. (2016). Device-associated infection and mortality rates, bacterial resistance, and length of stay in hospitals of Malaysia: International Nosocomial Infection Control Consortium (INICC)'s findings. *Canadian Journal of Infection Control Summer*, 31(2), 107–112. https://www.researchgate.net/publication/315114757\_Device-associated\_infection\_and\_mortality\_rates\_bacterial\_resistance\_and\_length\_of\_stay\_in\_ho spitals of Malaysia International Nosocomial Infection
- Results | Agency for Healthcare Research and Quality. (2017, November). Agency for Healthcare Research and Quality, Rockville, MD. https://www.ahrq.gov/hai/pfp/haccost2017-results.html
- Rosenthal, V. D., Duszynska, W., Ider, B. E., Gurskis, V., Al-Ruzzieh, M. A., Myatra, S. N., Gupta, D., Belkebir, S., Upadhyay, N., Zand, F., Todi, S. K., Kharbanda, M., Nair, P. K., Mishra, S., Chaparro, G., Mehta, Y., Zala, D., Janc, J., Aguirre-Avalos, G., ... Erben, N. (2021). International Nosocomial Infection Control Consortium (INICC) report, data summary of 45 countries for 2013-2018, Adult and Pediatric Units, Device-associated Module. *American Journal of Infection Control*, 49(10), 1267–1274. https://doi.org/10.1016/J.AJIC.2021.04.077
- Stevens, V., Geiger, K., Concannon, C., Nelson, R. E., Brown, J., & Dumyati, G. (2014). Inpatient costs, mortality and 30-day re-admission in patients with central-line-associated bloodstream infections. *Clinical Microbiology and Infection: The Official Publication of the European Society of Clinical Microbiology and Infectious Diseases*, 20(5). https://doi.org/10.1111/1469-0691.12407
- Sulong, A., Ramli, R., Canselor, H., & Mukhriz, T. (2013). Central line-associated blood stream infections: Surveillance and incidence in Intensive Care Unit at a Malaysian Medical Centre. *Malaysian Medical Centre*. *The Internet Journal of Infectious Diseases*, 12(2). https://www.researchgate.net/publication/250613577
- Tai, L. L., Lim, C. H., Mohd Nor, M. R., Ismail, N. I., & Wan Ismail, W. N. (2018).
  Malaysian Registry of Intensive Care Report for 2017. http://www.crc.gov.my/report-registry/
- Tan, C. C., Zanariah, Y., Lim, K. I., & Balan, S. (2007). Central Venous Catheter-Related Blood Stream Infections: Incidence and an Analysis of Risk Factors. *Med J Malaysia*, 62, 370–374. http://www.e-mjm.org/2007/v62n5/Central Venous Catheter.pdf

- Tarricone, R., Torbica, A., Franzetti, F., & Rosenthal, V. D. (2010). Hospital costs of central line-associated bloodstream infections and cost-effectiveness of closed vs. open infusion containers. The case of Intensive Care Units in Italy. *Cost Effectiveness and Resource Allocation*, 8(1), 1–10. https://doi.org/10.1186/1478-7547-8-8/TABLES/7
- Wang, H., Tong, H., Liu, H., Wang, Y., Wang, R., Gao, H., Yu, P., Lv, Y., Chen, S., Wang, G., Liu, M., Li, Y., Yu, K., & Wang, C. (2018). Effectiveness of antimicrobial-coated central venous catheters for preventing catheter-related blood-stream infections with the implementation of bundles: a systematic review and network meta-analysis. *Annals of Intensive Care*, 8(1), 71. https://doi.org/10.1186/S13613-018-0416-4
- Ziegler, M. J., Pellegrini, D. C., & Safdar, N. (2014). Attributable mortality of central line associated bloodstream infection: systematic review and meta-analysis. *Infection 2014* 43:1, 43(1), 29–36. https://doi.org/10.1007/S15010-014-0689-Y
- Zimlichman, E., Henderson, D., Tamir, O., Franz, C., Song, ; Peter, Yamin, C. K., Denham, C. R., & Bates, D. W. (2013). Health Care-Associated Infections A Meta-analysis of Costs and Financial Impact on the US Health Care System. *JAMA Intern Med*, 173(22), 2039–2046. https://doi.org/10.1001/jamainternmed.2013.9763